CLINICAL TRIAL: NCT02425371
Title: Optimized Management of Comorbidity in Heart Failure With Preserved Ejection Fraction in the Elderly (>60 Years) (OPTIMIZE-HFPEF)
Brief Title: Optimized Management of Comorbidity in Heart Failure With Preserved Ejection Fraction in the Elderly (>60 Years)
Acronym: OPTIMIZE-HFPEF
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Göteborg University (Other)
Collaborators: Umeå University (Other); Karolinska Institutet (Other); Uppsala University (Other); Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VGFOUREG-127071
Record Dates: First submitted 2015-02-25; First posted 2015-04-24 (Estimated); Last update posted 2018-09-07 (Actual); Status verified 2018-09

CONDITIONS: Heart Failure, Diastolic
MeSH Terms: conditions — Heart Failure, Diastolic | interventions — Mass Screening

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): screening and treatment of comorbidities
  Interventions: Other: Screening and treatment of comorbidities
- Control (Placebo Comparator): No screening of comorbidity
  Interventions: Other: Placebo Comparator

INTERVENTIONS:
Other: Screening and treatment of comorbidities — Screening and treatment of comorbidities
  Arms: Intervention
Other: Placebo Comparator — No screening of comorbidities
  Arms: Control

SUMMARY:
Growing recognition of the importance of co-morbidities in Heart Failure with Preserved Ejection Fraction (HFPEF) has led to the realization that rather than being a distinct disease entity, HFPEF may represent a spectrum of co-morbidities in elderly breathless patients. Accordingly, progress in managing HFPEF in the elderly requires improved understanding of HFPEF pathogenesis with a focus on the impact of co-morbidities. However, the available evidence is insufficient to determine the true prevalence and severity of co-morbidities as well as their impact on both diagnosis and treatment in HFPEF. Therefore there are widespread diagnostic uncertainty without proven therapy!

The purpose of this project is twofold:

1. The investigators will study how to improve diagnostic accuracy for HFPEF in elderly patients, despite frequent comorbidities and higher age? How useful is it to add exercise testing and contrast echocardiography as well as biomarker as additional diagnostic tools in elderly HFPEF patients?
2. The investigators will test the hypothesis that HFPEF in the elderly is dominated by multiple co-morbidities that are a major part of the syndrome itself that contribute to the development of HFPEF. This hypothesis implies that the treatment of co-morbidities will improve prognosis.

The investigators' overall goal is to bring about a paradigm shift in managing elderly patients with HFPEF by not only improving diagnosis but also effectively treating co-morbidities that are currently considered predisposing factors to HFPEF. This contrasts with trials during last two decades that only target the heart.

The investigators will pursue the following specific aims:

1. Validate the diagnostic criteria for HFPEF proposed by European Society of Cardiology 2012, and determine the added diagnostic values of exercise testing and contrast echocardiography as well as biomarker for HFPEF in a multi-center study.
2. Determine if systematic screening and optimal management of co-morbidities associated with HFPEF improves the outcomes of patients with HFPEF in a randomized study.

DETAILED DESCRIPTION:
Heart failure is primarily a disease of the elderly, with approximately half of these cases occurring in patients aged ≥75 years. Heart failure is the leading cause of hospitalization in the elderly. Moreover, it worsens cognition, physical function and quality of life, increases health care costs and leads to higher mortality. Nearly half of the patients with heart failure have preserved ejection fraction (HFPEF), and the prevalence appears to be rising. Although patterns of morbidity and functional decline are similar in patients with HFPEF to those with heart failure and reduced ejection fraction (HFREF), HFPEF represents a particular challenge since there is no proven treatment. Therapies that are effective in HFREF, including angiotensin-converting enzyme inhibitors, angiotensin receptor blockers and beta blockers, have so far been unsuccessful in HFPEF. This differential response to therapy combined with distinct patterns of structural remodeling suggests that HFPEF and HFREF are two discrete entities with fundamentally different pathophysiologies. A recently proposed mechanism for HFPEF development identifies a systemic pro-inflammatory state induced by comorbidities as the primary cause of HFPEF. Therefore, progress in managing HFPEF requires improved understanding of HFPEF pathogenesis with a focus on the impact of comorbidities.

Hypothesis: HFPEF in the elderly is dominated by multiple comorbidity which are not a complicating factor in HFPEF, but a major part of the syndrome, contribute to the HFPEF. Therefore, to make comorbidity as attractive therapeutic target will promote a paradigm shift toward individualized optimal care in elderly patients with HFPEF.

Main purpose: To promote a paradigm shift toward individualized optimal care in elderly patients with HFPEF by effective treatment of the comorbidities.

Specific aim: To determine if systematic screening and optimal management of comorbidities associated with HFPEF will improve outcome in patients with HFPEF

Work plan: The investigators' intervention study will use a multi-centre, prospective, randomized, open procedure but blinded end-point (PROBE) design. Patients (n=220) are randomized 1:1 to either usual care (n=110) or intervention (n=110). Inclusion criteria are HFPEF >60 years. In the Intervention arm, all patients will be subject to systematic screening and optimal treatment of 12 most frequently seen co-morbidity. Endpoints will be collected by Independent Endpoint Committee once a year during 2 years.

Significance and clinical relevance : The present study focuses on an important issue in the investigators' society, namely HFPEF in the elderly population. This health problem has been largely ignored despite the fact that there is no recommended therapy. The investigators' proposed study represents a paradigm shift in therapy. It is based on a new concept focusing on comorbidities that are considered to be predisposing factors to HFPEF in contrast to available trials that target only the heart. The investigators' study therefore challenges the current clinical practice and may fill the knowledge gap in HFPEF.

ELIGIBILITY:
Inclusion Criteria:

1. Validated HFPEF
2. Age >60 years
3. Chronic Heart Failure with at least one hospitalization or increased use of diuretics due to worsening is required during the last year
4. New York Heart Association class II -IV
5. Regarded as optimally treated and stable for at least 4 weeks (physician's opinion)

Exclusion Criteria:

1. Currently enrolled in another study
2. Significant chronic obstructive pulmonary disease (COPD) with forced expiratory volume within one second (FEV1) < 30% (European Respiratory Society criteria) in the last 4 weeks before randomization
3. Glomerular filtration rate (GFR) <30 ml/min/1.73m2 (Modification of Diet in Renal Disease [MDRD] GFR Equation)
4. Significant primary valve disease
5. Body mass index (BMI) >40
6. Severe cognitive dysfunction or dementia
7. Expected survival of less than one year
8. Planned cardiac surgery, Percutaneous Coronary Intervention

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 410 (Estimated)
Dates: Start 2014-09; Primary Completion 2019-03 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
A composite endpoint about which includes the patient's well-being symptoms (improved or worsened) | Change between baseline and after 2 years
  A composite endpoint about which includes the patient's well-being symptoms (improved or worsened). The endpoint consists of 4 effect categories composites that are determined on an individual basis at baseline and at 12 months. Each effect category has to meet either all 4 main criteria (1) Lickert scale 5 levels(breathlessness); (2) Lickert scale (tiredness); (3) NT-proBNP change of 30% from baseline; and (4) any events such the occurence of deaths mortality, hospital admission for heart failure or, use of intravenous diuretics during 12 months

SECONDARY OUTCOMES:
All cause mortality or hospitalization | Change between baseline and after 2 years
  All cause mortality or hospitalization due to cardiovascular causes (time to first event); All cause mortality;
  Total number of hospitalizations; The non-fatal clinical progression of heart failure, assessed subjectively by patients and physicians and objectively by the occurrence of major clinical events.

CONTACTS AND LOCATIONS:
Overall Officials: Michael X Fu, Professor, Principal Investigator — Göteborg University
Locations (1):
- Dept. Medicine, Gothenburg, Vastragotaland, Sweden

REFERENCES:
- [Background] Fu M, Zhou J, Thunstrom E, Almgren T, Grote L, Bollano E, Schaufelberger M, Johansson MC, Petzold M, Swedberg K, Andersson B. Optimizing the Management of Heart Failure With Preserved Ejection Fraction in the Elderly by Targeting Comorbidities (OPTIMIZE-HFPEF). J Card Fail. 2016 Jul;22(7):539-44. doi: 10.1016/j.cardfail.2016.01.011. Epub 2016 Jan 25. PMID 26820355